CLINICAL TRIAL: NCT06375759
Title: Subarachnoid-Subarachnoid (S-S) Bypass Versus Adhesion Lysis in Spinal Arachnoiditis and Syringomyelia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XWSSB
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Syringomyelia
Keywords: syringomyelia
MeSH Terms: conditions — Syringomyelia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subarachnoid-Subarachnoid (S-S) Bypass (Experimental): After dissections of the normal arachnoid mater at the cephalic and caudal sites, 1 or 2 tubes made of medical grade silicone (ventricular drainage tube; internal diameter 1.5-2.0 mm, external diameter 2.5-3.3 mm) were inserted into the cephalic and caudal ends of the normal subarachnoid space. The part of the tube inserted into the subarachnoid space was approximately 2 cm long. The total length of the tube was equal to the distance between the cephalic and caudal ends of the normal dissected arachnoid mater, along with approximately 4 cm of extra tubing.
  Interventions: Procedure: Subarachnoid-Subarachnoid (S-S) Bypass
- Intradural Adhesion Lysis (Active Comparator): The dura is opened sharply, exposing the spinal cord. After microsurgical dissection adhesion, the dura is sewn closed with a dural graft.
  Interventions: Procedure: Intradural Adhesion Lysis

INTERVENTIONS:
Procedure: Subarachnoid-Subarachnoid (S-S) Bypass — The dura was widely exposed beyond the level of trauma, and then a midline dural opening was made under an operative microscope. When dura and arachnoid were adhered because of an expansion of arachnoiditis, they had to be released with great care to place the bypass tubes. During this procedure, S-S bypass was not usually needed to performed arachnoid lysis. This exposure had to reach the normal arachnoid mater free from arachnoiditis and adhesion, with normal CSF circulation.
  After dissections of the normal arachnoid mater at the cephalic and caudal sites, 1 or 2 tubes made of medical grade silicone (ventricular drainage tube; internal diameter 1.5-2.0 mm, external diameter 2.5-3.3 mm) were inserted into the cephalic and caudal ends of the normal subarachnoid space. The part of the tube inserted into the subarachnoid space was approximately 2 cm long.
  Arms: Subarachnoid-Subarachnoid (S-S) Bypass
Procedure: Intradural Adhesion Lysis — Intradural spinal cord Adhesion Lysis
  Arms: Intradural Adhesion Lysis

SUMMARY:
To determine whether Subarachnoid-Subarachnoid (S-S) Bypass results in better patient outcomes with fewer complications and improved quality of life compared to intradural adhesion lysis in individuals with Spinal Arachnoiditis and Syringomyelia.

DETAILED DESCRIPTION:
Participants with Spinal Arachnoiditis and Syringomyelia will be randomized to either have a Subarachnoid-Subarachnoid (S-S) Bypass or intradural adhesion Lysis. The participant will then return to the neurosurgeon's office at the following time points which are consistent with standard of care practice: 3-6 months, 12 and 24 months. At these visits, the clinician will complete a physical exam and the participant will report on the prognosis of symptoms and complete questionnaires. A spine MRI will be performed 3-6 months, 12 and 24 months after the decompression.

ELIGIBILITY:
Inclusion Criteria:

* 1) history of traumatic spinal cord injury or other infection; 2) evidence of progressive neurological deficit, and/or pain syndrome; 3) MRI showing a syringomyelia due to spinal trauma or other infection; and 4) minimum follow-up period of more than 1 year.

Exclusion Criteria:

* Chiari-malformation, myelomalacia, subarachnoid cyst, syringomyelia due to other spinal diseases (such as degenerative spinal disease)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
complication | 12 months
  Reoperation,Wound infection,Aseptic meningitis,CSF fistula,Subcutaneous hydrops,Other complications

SECONDARY OUTCOMES:
improvement or resolution of the syrinx, | 3-6, 12 and 24 months
  defined as > 50% improvement in length, maximal cross-sectional diameter, or both.
ASIA score | 3-6, 12 and 24 months
  American Spinal Injury Association(ASIA) Score for evaluating the spinal cord function， degree of the spinal cord function, motor1-100, sensory 1-224, higher scores mean a better outcome
Klekamp and Sammi syringomyelia scale | 3-6, 12 and 24 months
  for evaluating the spinal cord function, higher scores mean a better outcome
modified Japanese Orthopaedic Association Scores (mJOA) | 3-6, 12 and 24 months
  Motor function， sensory， bladder function；for evaluating the spinal cord function；0-17， higher scores mean a better outcome
xuanwu syringomyelia scale | 3-6, 12 and 24 months
  for evaluating the spinal cord function, for evaluating the spinal cord function；0-18， higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Fengzeng Jian, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Hayashi T, Ueta T, Kubo M, Maeda T, Shiba K. Subarachnoid-subarachnoid bypass: a new surgical technique for posttraumatic syringomyelia. J Neurosurg Spine. 2013 Apr;18(4):382-7. doi: 10.3171/2013.1.SPINE12828. Epub 2013 Feb 22. PMID 23432327
- [Background] Heiss JD. Cerebrospinal Fluid Hydrodynamics in Chiari I Malformation and Syringomyelia: Modeling Pathophysiology. Neurosurg Clin N Am. 2023 Jan;34(1):81-90. doi: 10.1016/j.nec.2022.08.007. Epub 2022 Nov 3. PMID 36424067
- [Background] Hemley SJ, Bilston LE, Cheng S, Stoodley MA. Aquaporin-4 expression and blood-spinal cord barrier permeability in canalicular syringomyelia. J Neurosurg Spine. 2012 Dec;17(6):602-12. doi: 10.3171/2012.9.SPINE1265. Epub 2012 Oct 19. PMID 23082850
- [Background] Guan J, Yuan C, Yao Q, Du Y, Fang Z, Zhang L, Jia S, Zhang C, Liu Z, Wang K, Duan W, Wang Z, Wang X, Wu H, Chen Z, Jian F. A novel scoring system for assessing adult syringomyelia associated with CM I treatment outcomes. Acta Neurol Belg. 2023 Jun;123(3):807-814. doi: 10.1007/s13760-023-02264-4. Epub 2023 Apr 12. PMID 37046133
- [Background] Guan J, Yuan C, Zhang C, Ma L, Yao Q, Cheng L, Liu Z, Wang K, Duan W, Wang X, Wu H, Chen Z, Jian F. Intradural Pathology Causing Cerebrospinal Fluid Obstruction in Syringomyelia and Effectiveness of Foramen Magnum and Foramen of Magendie Dredging Treatment. World Neurosurg. 2020 Dec;144:e178-e188. doi: 10.1016/j.wneu.2020.08.068. Epub 2020 Aug 15. PMID 32805463
- [Result] Yuan C, Xia P, Duan W, Wang J, Guan J, Du Y, Zhang C, Liu Z, Wang K, Wang Z, Wang X, Wu H, Chen Z, Jian F. Long-Term Impairment of the Blood-Spinal Cord Barrier in Patients With Post-Traumatic Syringomyelia and its Effect on Prognosis. Spine (Phila Pa 1976). 2024 Mar 15;49(6):E62-E71. doi: 10.1097/BRS.0000000000004884. Epub 2023 Nov 28. PMID 38014747